CLINICAL TRIAL: NCT06805539
Title: Decentralised Observational Disease Area Study Exploring Remote Collection of Data in Adult Participants With Overweight Condition or Obesity Undergoing Weight Management Program
Brief Title: A Study Collecting Remote Data in People With an Overweight Condition or Obesity on a Weight Management Program
Status: Active, not recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-7632; U1111-1301-4301 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Overweight, Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consent video: Participants watching a pre-recorded consent video.
  Interventions: Other: No treatment given
- Video call: Participants obtaining the information regarding the study at a video call from the study staff.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this study is to collect health data related from participants living with an overweight condition in a decentralised clinical study set-up. All data will be collected remotely using an app downloaded on your personal smartphone and devices (watch and scale).

Participants will participate in this study for 24 weeks. The study does not include any study medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Informed electronic consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Willingness to consent via the e-consent process before any study-related activities (study- related activities are any procedure related to recording of data according to the protocol)
3. Male or female, age above or equal to 18 years at the time of signing informed consent
4. Body mass index (BMI) above or equal to 25 kg/m^2 self-reported in the Confirmation of Eligibility Questionnaire
5. About to initiate/has initiated at least one of the following weight management program(s) :

   1. Diet regime aimed at losing weight and/or
   2. Exercise regime aimed at losing weight and/or
   3. Prescription of any approved anti-obesity medication (according to standard practice) as prescribed by the participant's treating physician
6. Willingness to follow study procedures
7. Willingness to, and capable of using the study devices and app
8. Fluent in oral and written Danish language
9. In possession of a compatible smartphone (minimum Android 10 and iOS14) throughout the study that has a reliable internet connection, regular connection to 4G/5G network, or Wi-Fi and that has the capability of downloading the study app and connecting with the smartwatch, the body composition scale and the data hub)

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Participation in any study investigating an overweight condition or obesity
3. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
4. Type 1 or type 2 diabetes
5. Currently under treatment with any GLP-1 RA with the indication of improving glycaemic control
6. Currently using a pacemaker, an implantable cardioverter-defibrillator (ICD) or cardiac resynchronisation therapy (CRT) due to the electrical effects of the body composition scale
7. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an effective contraceptive method during the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with an overweight condition or obesity undergoing weight management prescribed by a general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion of the electronic informed consent process (e-consent) | Week -2 to week 0
  Count
Body weight measurements recorded | From week 0 (device set-up date) to the week 24 (end of study)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk committment on novonordisk-trials.com
URL: https://novonordisk-trials.com